CLINICAL TRIAL: NCT00185068
Title: A Prospective, Open Label, Titration Study to Assess the Efficacy and Safety of Benicar® and Benicar ®HCT in Patients With Stage II Systolic Hypertension
Brief Title: An Examination of the Safety and Blood Pressure Lowering Effect of Increasing Doses of Benicar® and Benicar® HCT in Patients With Hypertension
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Daiichi Sankyo (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 866-443
Record Dates: First submitted 2005-09-09; First posted 2005-09-16 (Estimated); Last update posted 2005-09-16 (Estimated); Status verified 2005-09

CONDITIONS: Hypertension
Keywords: Systolic hypertension, Angiotensin receptor blocker
MeSH Terms: conditions — Hypertension; Isolated Systolic Hypertension | interventions — Olmesartan Medoxomil; Hydrochlorothiazide

INTERVENTIONS:
Drug: Olmesartan medoxomil
Drug: Olmesartan medoxomil/hydrochlorothiazide
Drug: Hydrochlorothiazide

SUMMARY:
Effect of increasing doses of olmesartan medoxomil and olmesartan medoxomil/hydrochlorothiazide on blood pressure in patients with hypertension

ELIGIBILITY:
Inclusion Criteria:

* 1. 18 years of age.
* 2. Patients with stage II systolic hypertension
* 3. If female, must have negative serum pregnancy test at screening and be either post-menopausal, had a hysterectomy or tubal ligation at least 6 months before consent or if of childbearing potential, must practice approved measures of birth control throughout study.

Exclusion Criteria:

* 1. Hypertensive encephalopathy, stroke or transient ischemic attack (TIA) within the past 6 months.

  2. History of myocardial infarction, percutaneous transluminal coronary revascularization, coronary artery bypass graft, and/or unstable angina pectoris within the past 6 months.

  3. Severe hypertension (DBP greater than or equal to 110 mm Hg or SBP > 200 mm Hg).

  4. History of secondary hypertension including renal disease, phaeochromocytoma, or Cushing's disease.

  5. Type I diabetes mellitus. 6. Evidence of symptomatic resting bradycardia, congestive heart failure, or hemodynamically significant cardiac valvular disease.

  7. Presence of heart block greater than first degree sinoatrial block, Wolff-Parkinson-White Syndrome, Sick Sinus Syndrome, Atrial fibrillation, or Atrial Flutter.

  8. Laboratory test values considered clinically significant by the investigator.

  9. Evidence of liver disease as indicated by SGOT or SGPT and/or total bilirubin > 3 times the upper limit of normal.

  10. Pregnant or lactating females.
* 11. Patients with malignancy during the past 5 years excluding squamous cell or basal cell carcinoma of the skin.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110
Dates: Start 2004-03; Study Completion 2004-10

PRIMARY OUTCOMES:
Change in mean trough seated systolic blood pressure compared to the start of the study

SECONDARY OUTCOMES:
1. Blood pressure changes from baseline at the end of each titration period.
2. Percentage of patients responding to therapy
3. Percentage of patients achieving various blood pressure target goals

CONTACTS AND LOCATIONS:
Locations (16):
- United States (16):
  - Fort Lauderdale, California
  - Long Beach, California
  - Roseville, California
  - Sacramento, California
  - Santa Anna, California
  - Tustin, California
  - Westlake Village, California
  - DeLand, Florida
  - Pembroke Pines, Florida
  - Orland Park, Illinois
  - New Orleans, Louisiana
  - Auburn, Maine
  - Omaha, Nebraska
  - Buffalo, New York
  - Oklahoma City, Oklahoma
  - Madison, Wisconsin